CLINICAL TRIAL: NCT04986059
Title: Effects of Pre-event Massage on Muscle Activity During Jump Activities on Gastrocnemius and Hamstring Muscles
Brief Title: Effects of Pre-event Massage on Muscle Activity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Albert Pérez Bellmunt, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol 4B
Record Dates: First submitted 2021-07-22; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Neuromuscular Diseases
Keywords: Pre-competition massage; Pre-event massage; Gastrocnemius; Superficial Electromyography; Hamstrings
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-event massage (Experimental)
  Interventions: Other: Pre-event massage
- Control (No Intervention)

INTERVENTIONS:
Other: Pre-event massage — Five minutes massage, combining superficial and high-frequency techniques of massage applied with the therapist hands on gastrocnemius and hamstring muscles
  Arms: Pre-event massage

SUMMARY:
The study observes the effect of a pre-event massage on the gastrocnemius and Hamstring muscles on muscle activity.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Muscle injury in the last two months
* Suffer a musculoskeletal disorder that doesn't allow the subject to do the study protocol

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Muscle activity (microVolts) | Change between baseline(immediately before intervention) and post intervention (immediately after intervention
  sEMG is a NON-invasive method that measures the electrical activity of the muscle generated by the passage of the nerve impulse, which causes depolarization of the muscle cell membrane during excitation. Once the muscle is contracted and receives electrical signals, the electrodes pick up these signals and record them on the device application.

SECONDARY OUTCOMES:
Jump Force (Newtons) | Change between baseline(immediately before intervention) and post intervention (immediately after intervention)
  Jump Force will be measured using the Myjump app
Jump speed (m/s) | Change between baseline(immediately before intervention) and post intervention (immediately after intervention)
  Jump Speed will be measured using the Myjump app
Jump Height (cm) | Change between baseline(immediately before intervention) and post intervention (immediately after intervention)
  Jump Height will be measured using the Myjump app

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional Catalunya, Barcelona, Sant Cugat, Spain